CLINICAL TRIAL: NCT06604026
Title: An Investigational Study to Evaluate the Safety and Performance of the BD PosiFlush™ SafeScrub on Needleless Access Devices
Brief Title: Investigational Study With the BD PosiFlush™ SafeScrub on NADs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MDS-23PFINTEU001
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-05

CONDITIONS: CRBSI - Catheter Related Bloodstream Infection

STUDY DESIGN:
Intervention Model Description: At each participating site, one medical or surgical unit will conduct the treatment arm and one unit will conduct the control arm randomizing which unit will perform the treatment or control arm at the study site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): use of the BD PosiFlush™ SafeScrub device
  Interventions: Device: BD PosiFlush™ SafeScrub
- Control Arm (Active Comparator): pre-filled saline syringe (BD PosiFlush™ SP Syringe) and alcohol pad
  Interventions: Device: BD PosiFlush™

INTERVENTIONS:
Device: BD PosiFlush™ SafeScrub — Clinicians will be advised to use BD PosiFlush™ SafeScrub as per the Instructions for Use for the treatment arm of the study.
  An independent nurse observer will observe and document any adverse events (e.g.
  local skin reaction, or irritation, or allergic response, up to and including symptoms of anaphylaxis), compliance with needleless access device scrubbing before flushing, device success rate (encapsulation and removal) as well as the time requirements and number of steps for needleless access device scrubbing prior to catheter flushes during medication administration process.
  Arms: Treatment arm
Device: BD PosiFlush™ — Clinicians will be advised to follow and document the respective unit protocol, while using the standard pre-filled syringe (BD PosiFlush™ SP Syringe) and alcohol pad for scrubbing and flushing of NADs in the control arm of the study as the routine practice.
  An independent nurse observer will observe and document any adverse events (e.g.
  local skin reaction, or irritation, or allergic response, up to and including symptoms of anaphylaxis), compliance with needleless access device scrubbing before flushing, device success rate (encapsulation and removal) as well as the time requirements and number of steps for needleless access device scrubbing prior to catheter flushes during medication administration process.
  Arms: Control Arm

SUMMARY:
This study is an investigational study to evaluate the safety and performance of the BD PosiFlush™ SafeScrub on needleless access devices.

DETAILED DESCRIPTION:
This study is being conducted to generate clinical data to support the performance and safety of BD PosiFlush™ SafeScrub. The study data will be used for regulatory submission in EU.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient (≥18 years of age) in a high acuity hospital medical or surgical unit regardless of gender, with an eligible in-situ vascular access device and with a needleless access device (NAD). This includes patients who have a current VAD, whether it is newly placed or long-term access as part of their routine medical care. Eligible in-situ vascular access devices are peripheral intravenous catheters (PIVCs), peripherally inserted central catheters (PICCs), central venous catheters (CVCs) and implanted venous access ports. Eligible NADs are stopcocks, Y-sites, and needle-free connectors.
2. Expected to be available until 2 accesses are completed and for any periodic observation upto 15 min after each access.
3. Able and willing to provide informed consent or legal authorized representative (LAR) authorized to give consent on behalf of the participant.

Exclusion Criteria:

Any patient in whom observation might interfere with medical care or create undue hardship as determined by the patients care team.

* Patients under the age of 18.
* Patients suffering hypernatremia and fluid retention, when the administration of sodium or chloride could be clinically detrimental as determined by the study investigator.
* Patients with a known allergy to any of the followings as determined by the study investigator:
* Any of the components or materials of BD PosiFlush™ SafeScrub device or BD PosiFlush™ SP Syringe, or
* 0.9% sodium chloride solution
* Pregnant or breastfeeding women
* Urine pregnancy test will be required for all women of childbearing age who want to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Device related adverse events | 15 minutes
  To assess the incidence of BD PosiFlush™ SafeScrub device-related adverse events up to 15 min after each access

SECONDARY OUTCOMES:
Compliance rate of device scrubbing | 15 minutes
  To assess if the compliance rate of needleless access device scrubbing before flushing with use of BD PosiFlush™ SafeScrub is higher compared to standard practice (i.e., use of pre-filled syringe (BD PosiFlush™ SP Syringe) and an alcohol pad) up to 15 min after each access
Device success rate | 15 minutes
  To assess the performance of the BD PosiFlush™ SafeScrub. Percent success rate (≥85%) for BD PosiFlush™ SafeScrub to encapsulate the needleless access device, and to be removed from the needleless access device up to 15 min after each access

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Van Laethem, Study Chair — Becton, Dickinson and Company BD Medication Delivery Systems/Catheter Care
Locations (2):
- Austria (2):
  - Ordensklinikum Linz Elisabethinen, Linz, Upper Austria
  - Medical University Vienna, Vienna

IPD SHARING:
Plan to Share IPD: No